CLINICAL TRIAL: NCT04527029
Title: The Studies of Early Intelligent Diagnosis of Limb Deformity in Children by AI and Clinic Application
Brief Title: Early Intelligent Diagnosis of Limb Deformity in Children by AI and Clinic Application
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ningbo1528
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Limb Deformity
Keywords: Limb deformity; Pediatrics ; Artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- limb deformity children: the imaging of limb deformity diagnosis by AI
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — It is an observational study. No interventions.

SUMMARY:
The limb deformity in children include congenital limb malformations or acquired from the damage of epiphyseal plate which caused by tumor, inflammation and trauma. Due to the complexity of the disease itself, rapid dynamic development and the characteristics of children's growth and development, the deformities are constantly changing. In addition, the serious lack of clinical diagnosis and treatment resources in the Department of Pediatric Orthopedics has led to the misdiagnosis and improper treatment of children's limb deformities. Thus, its necessary to find an intelligent way to help doctor to early diagnosis of limb deformity and provide a proper treatment in children.

DETAILED DESCRIPTION:
The extraction and application of big data of children's limb deformities, intelligent labeling of image data, precise positioning, and perfecting the anatomical data of children's limb deformities.Improve the positioning accuracy of key points in X-ray images of children's limb deformities by means of step-by-step supervision to improve the accuracy of diagnosis.Realize an intelligent report generation system that combines patient background information, establish an end-to-end auxiliary diagnosis and treatment suggestion demonstration application system; realize a full set of artificial intelligence solutions for children's skeletal deformities, early screening and diagnosis of children, and forming an intelligent referral system of children's limb deformities.

ELIGIBILITY:
Inclusion Criteria:

Children with limb deformity

Exclusion Criteria:

Children without limb deformity

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with limb deformity
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Deformity detection | At enrollment
  It is a binary variable (1/0). The radiographic features of children would be evaluated by artificial Intelligence. If the deformity was detected, variable would be setted into 1.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ning, PhD, Principal Investigator — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirskaia NB, Kolomenskaia AN, Siniakina AD. [Prevalence and medical and social importance of disorders and diseases of the musculoskeletal systems in children and adolescents (review of literature)]. Gig Sanit. 2015 Jan-Feb;94(1):97-104. Russian. PMID 26031051
- [Background] Theofilatos K, Pavlopoulou N, Papasavvas C, Likothanassis S, Dimitrakopoulos C, Georgopoulos E, Moschopoulos C, Mavroudi S. Predicting protein complexes from weighted protein-protein interaction graphs with a novel unsupervised methodology: Evolutionary enhanced Markov clustering. Artif Intell Med. 2015 Mar;63(3):181-9. doi: 10.1016/j.artmed.2014.12.012. Epub 2015 Feb 18. PMID 25765008
- [Background] Silverman BG, Hanrahan N, Bharathy G, Gordon K, Johnson D. A systems approach to healthcare: agent-based modeling, community mental health, and population well-being. Artif Intell Med. 2015 Feb;63(2):61-71. doi: 10.1016/j.artmed.2014.08.006. Epub 2014 Sep 11. PMID 25801593
- [Background] Jamaludin A, Lootus M, Kadir T, Zisserman A, Urban J, Battie MC, Fairbank J, McCall I; Genodisc Consortium. ISSLS PRIZE IN BIOENGINEERING SCIENCE 2017: Automation of reading of radiological features from magnetic resonance images (MRIs) of the lumbar spine without human intervention is comparable with an expert radiologist. Eur Spine J. 2017 May;26(5):1374-1383. doi: 10.1007/s00586-017-4956-3. Epub 2017 Feb 6. PMID 28168339
- [Background] Ravi D, Wong C, Deligianni F, Berthelot M, Andreu-Perez J, Lo B, Yang GZ. Deep Learning for Health Informatics. IEEE J Biomed Health Inform. 2017 Jan;21(1):4-21. doi: 10.1109/JBHI.2016.2636665. Epub 2016 Dec 29. PMID 28055930
- [Background] Rahmathulla G, Nottmeier EW, Pirris SM, Deen HG, Pichelmann MA. Intraoperative image-guided spinal navigation: technical pitfalls and their avoidance. Neurosurg Focus. 2014 Mar;36(3):E3. doi: 10.3171/2014.1.FOCUS13516. PMID 24580004